CLINICAL TRIAL: NCT03155672
Title: A PHASE I, SINGLE-CENTER, MIXED METHODS STUDY ON THE HEALTH OUTCOMES OF VISUAL SELF EXPRESSION
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 01017
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: A Healthcare Professional, a Patient or Caregiver in the Radiation Oncology Department at the University of Pennsylvania
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Art therapy — Art Therapy

SUMMARY:
To gain understanding about the impact of visual art making on biomarkers, such as cortisol, alpha amylase, oxytocin, etc. to examine whether and to what extent there are changes in levels of stress and immune function in patients and caregivers adults (including family caregivers and medical professionals)

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 18 - 70
* A healthcare professional, a patient or caregiver in the Radiation Oncology Department at the University of Pennsylvania
* Subjects must be capable of giving informed consent

Exclusion Criteria:

* Any healthcare professional or patient/caregiver not working in or being seen at Radiation Oncology Department at the University of Pennsylvania

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A healthcare professional, a patient or caregiver in the Radiation Oncology Department at the University of Pennsylvania
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
NUmber of changes in levels of stress and immune function in patients and caregivers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Levin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States